CLINICAL TRIAL: NCT06782295
Title: A Prospective Randomized Controlled Trial Comparing Constrained Condylar vs Posterior Stabilized Articulations in Revision Total Knee Arthroplasty
Brief Title: The Use of CCK vs PS in Revision TKAs
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Omar Behery, Principle Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25010208
Record Dates: First submitted 2025-01-03; First posted 2025-01-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Aseptic Loosening of Prosthetic Joint; Instability of Prosthetic Joint; Reimplantation for Periprosthetic Joint Infection; Femoral Revision Indicated; Tibial Component Revision
Keywords: revision total knee replacement; cck; ps; coronal instability; sagittal instability

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups: constrained condylar (CCK) vs posterior stabilized (PS) articulating bearings. These are standard bearings used in revision knees, comparing two types.
Masking Description: only the patient is blinded ahead of time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Constrained condylar (CCK) (Active Comparator): Once patient meets inclusion criteria, they'll be randomized prior to surgery to a specific CCK implant design. All surgeries will be done at the approved hospital or ASC and if the allocated component isn't used, the patient will still be followed post operatively and remain in the study.
  Interventions: Device: Constrained Condylar bearing
- Posterior Stabilized (PS) bearing (Active Comparator): Once patient meets inclusion criteria, they'll be randomized prior to surgery to a specific PS implant design. All surgeries will be done at the approved hospital or ASC and if the allocated component isn't used, the patient will still be followed post operatively and remain in the study.
  Interventions: Device: posterior stabilized bearing

INTERVENTIONS:
Device: Constrained Condylar bearing — Patients in this intervention will receive a CCK bearing component
  Other Names: CCK
  Arms: Constrained condylar (CCK)
Device: posterior stabilized bearing — Patients in this intervention will receive a PS bearing component
  Arms: Posterior Stabilized (PS) bearing

SUMMARY:
This study aims to compare the clinical impact of Constrained Condylar versus Posterior Stabilized Knee (PS) bearings on patient satisfaction and surgical outcomes including mid-term survivorship among patients undergoing revision total knee arthroplasty.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether a difference exists in clinical patient reported outcomes between CCK or PS bearings following rTKA. A secondary goal of the study is to compare both bearings in survivorship free of revision surgery as well as other surgical complications including instability, in early to mid-term follow-up.

ELIGIBILITY:
Inclusion criteria:

* Patients between 18-80 years of age
* Patients who are undergoing both femoral and tibial component revisions, or isolated femoral component revisions with a retained tibial component that is compatible with PS or CCK bearings
* Patients who are at least 6-weeks out from primary TKA surgery, with complete pre-operative and post-operative knee radiographs obtained at standard of care perioperative visits (AP/lateral and patellar views)
* Patients undergoing rTKA for indications including aseptic component loosening, flexion or extension coronal or sagittal instability, component malalignment, arthrofibrosis, patellar maltracking, reimplantation following single or two-stage exchange revision for prosthetic joint infection or bearing surface wear when femoral or tibial component revision is indicated.
* The use of revision total knee arthroplasty systems which have PS and CCK bearing options including different degree options of coronal and rotational constraint (to be individually randomized per constrained option):
* Zimmer Biomet Persona, NexGen, or Vanguard
* Smith and Nephew Legion
* DJO / Enovis Empowr
* Stryker Triathlon
* Link SymphoKnee
* Depuy Attune sion Criteria:

Exclusion Criteria:

Patients undergoing rTKA with a hinged implant, or pre-operatively determined to require CCK bearing rTKA, > 80 years of age, or those requiring rTKA less than 6-weeks from the primary TKA,

Patients undergoing rTKA for bearing exchange only rTKA, isolated tibial component rTKA

Patients with pre-operative diagnosis of extensor mechanism disruption or collateral ligament incompetence or with a compromised soft tissue envelope requiring pre-pre-operative plastic surgery evaluation and planned soft tissue coverage.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2038-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical patient reported outcomes | 6 weeks post op
  patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time. The clinical patient reported outcomes of a revision total knee replacement to detect a 6-point difference in knee society score (KSS)
Clinical patient reported outcomes | 1 year post op
  Patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time. The clinical patient reported outcomes of a revision total knee replacement to detect a 6-point difference in knee society score (KSS)
Clinical patient reported outcomes | 2 year post op
  Patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time. The clinical patient reported outcomes of a revision total knee replacement to detect a 6-point difference in knee society score (KSS)
Clinical patient reported outcomes | 5 year post op
  Patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time. The clinical patient reported outcomes of a revision total knee replacement to detect a 6-point difference in knee society score (KSS)
Clinical patient reported outcomes | 10 year post op
  Patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time. The clinical patient reported outcomes of a revision total knee replacement to detect a 6-point difference in knee society score (KSS)
Clinical patient reported outcomes | 20 year post op
  Patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time. The clinical patient reported outcomes of a revision total knee replacement to detect a 6-point difference in knee society score (KSS)

SECONDARY OUTCOMES:
Clinical reported outcomes (Koos Jr) | 6 weeks to 20 years post op
  patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time
Range of motion over time | pre op to 20 years pots op
  Patients will have their knee range of motion (ROM) checked prior to revision surgery and at multiple timepoints after surgery
Clinical reported outcomes ( VR-12) | 6 weeks, 1 year, 2 years, 5 years, 10 years, 15 years, 20 years post op
  patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time
Clinical reported outcomes ( Forgotten Joint Score) | 6 weeks to 20 years post op
  patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time
Clinical reported outcomes (EQ-5D-3L) | 6 weeks, 1 year, 2 years, 5 years, 10 years, 15 years, 20 years post op
  patients will be asked pre and post operatively to completed standard of care patient reported outcomes to compare over time

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No